CLINICAL TRIAL: NCT05269641
Title: The Effect of Almond Supplementation on Mild to Moderate Acne
Brief Title: Almond Supplementation on Mild to Moderate Acne
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Almond Board of California (Other)
Responsible Party: Principal Investigator, Raja Sivamani, MD MS AP, Principal Investigator, Integrative Skin Science and Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlmondAcne_01
Record Dates: First submitted 2022-02-12; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Acne Vulgaris
Keywords: microbiome; nutrition
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almonds (Experimental): Daily consumption of almonds.
  Interventions: Other: Food: whole almonds
- Control Snack (Placebo Comparator): Daily non-nut snack will be consumed.
  Interventions: Other: Food: non-nut snack

INTERVENTIONS:
Other: Food: whole almonds — 60g of whole almonds will be consumed daily.
  Arms: Almonds
Other: Food: non-nut snack — A non-nut snack will be consumed daily.
  Arms: Control Snack

SUMMARY:
This study will assess the effect of almond supplementation on acne and on gut health.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 15 years of age until 45 years of age.
* The presence of mild to moderate acne based on investigator global assessment.
* Individuals who have remained stable on their topical or oral acne regimen for at least 4 weeks, except if the medication is a noted exclusion.

Exclusion Criteria:

* The presence of severe acne as noted by the investigator global assessment.
* Those with a nut allergy.
* Those who are unwilling to discontinue oral probiotic-based supplementation to meet the washout criteria prior to enrolling.
* Those who are unwilling to discontinue topical antibiotics and topical benzoyl peroxide to meet the washout criteria prior to enrolling.
* Individuals who are unwilling to discontinue vitamin E containing supplements during the washout and intervention.
* Individuals who have been on an oral antibiotic for acne within the previous 1 month.
* Individuals who are pregnant or breastfeeding.
* Individuals who have changed any of their hormonal based contraception within 3 months prior to joining the study.
* Oral supplementation that has nuts in it.
* Use of isotretinoin within the three months prior to joining the study.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Total lesion count | 20 weeks
  Number of of inflammatory lesions, and open and closed comedones

SECONDARY OUTCOMES:
Inflammatory lesion count | 12 weeks
  Number of inflammatory lesions
Inflammatory lesion count | 20 weeks
  Number of inflammatory lesions
Non-inflammatory lesion count | 12 weeks
  Number of open and closed comedones
Non-inflammatory lesion count | 20 weeks
  Number of open and closed comedones
Investigator global assessment (IGA) of acne | 12 weeks
  Validated scale for global assessment of acne. Scale of 0-4, 4 indicating greater severity.
Investigator global assessment (IGA) of acne | 20 weeks
  Validated scale for global assessment of acne. Scale of 0-4, 4 indicating greater severity.
Quality of Life Survey | 12 weeks
  Dermatology quality of life index survey assessment (DQLI). Scale is 0 to 30, the higher the score the greater impairments to quality of life.
Quality of Life Survey | 20 weeks
  Dermatology quality of life index survey assessment (DQLI). Scale is 0 to 30, the higher the score the greater impairments to quality of life.
Sebum excretion | 12 weeks
  Measure of skin sebum via sebumeter.
Sebum excretion | 20 weeks
  Measure of skin sebum via sebumeter
Gut microbiome assessment | 12 weeks
  Gut microbiome shift for short-chain fatty acid producing bacteria via stool sample
Gut microbiome assessment | 20 weeks
  Gut microbiome shift for short-chain fatty acid producing bacteria via stool sample
Skin microbiome diversity | 12 weeks
  Shift in the Shannon diversity of the skin microbiome through adhesive strip and swab collection.
Skin microbiome diversity | 20 weeks
  Shift in the Shannon diversity of the skin microbiome through adhesive strip and swab collection.

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No